CLINICAL TRIAL: NCT01654692
Title: A Phase II Study of the Combination of Ipilimumab and Fotemustine in Patients With Unresectable Locally Advanced or Metastatic Malignant Melanoma
Brief Title: A Combination of Ipilimumab and Fotemustine for Treat Unresectable Locally Advanced or Metastatic Melanoma
Acronym: NIBIT-M1
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Italian Network for Tumor Biotherapy (Other)
Collaborators: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NIBIT-M1; 2010-019356-50 (EudraCT Number)
Record Dates: First submitted 2012-07-18; First posted 2012-08-01 (Estimated); Last update posted 2015-05-13 (Estimated); Status verified 2015-05

CONDITIONS: Metastatic Malignant Melanoma
Keywords: metastatic melanoma; Ipilimumab
MeSH Terms: conditions — Melanoma | interventions — Ipilimumab; fotemustine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Single arm of ipilimumab and fotemustine (Experimental): Ipilimumab in combination with Fotemustine
  Interventions: Drug: Ipilimumab and Fotemustine

INTERVENTIONS:
Drug: Ipilimumab and Fotemustine — Ipilimumab: 10 mg/kg q3 weeks for 4 doses, q12 weeks starting at Week 24 Fotemustine: 100 mg/m2 q1 week for 3 doses, q3 weeks starting at Week 9
  Other Names: Ipilimumab (Yervoy); Fotemustine (Muphoran)

SUMMARY:
This study is designed to assess the safety and efficacy of a combination of ipilimumab and fotemustine in Patients with Unresectable Locally Advanced or Metastatic Malignant Melanoma.

DETAILED DESCRIPTION:
Immunotherapy, chemotherapy and chemotherapy combinations are currently the most effective accepted systemic treatments for metastatic melanoma. However, significant and prolonged responses are rare.

The trial will determine the additional benefit achieved from adding fotemustine to the anti-CTLA-4 monoclonal antibody,ipilimumab .

It is assumed that the mechanism by which ipilimumab augments the effects of chemotherapy in animal models relies on the ability of the cytotoxic agent to induce apoptosis of tumor cells. These apoptotic cells then can function as potent inducers of an immune response against any non-tolerized antigen that they contain. Thus, the chemotherapy may be creating an in vivo autologous tumor vaccine. Ipilimumab prevents the down regulation of this immune response, allowing for tumor rejection. Animal models evaluating the combination of anti-CTLA4 antibody and chemotherapy have given only a brief acute treatment with chemotherapy - presumably adequate to induce some tumor apoptosis, but inadequate to induce significant prolonged tumor rejection.

Since patients with metastatic melanoma generally require therapy within a relatively short period of time, this protocol will allow for the use of fotemustine. Standard dosing of fotemustine will be used to optimize the chance for tumor control.

ELIGIBILITY:
Inclusion Criteria:

* Histologic diagnosis of malignant melanoma
* Stage III (unresectable) or Stage IV melanoma
* Maximum 1 line of chemotherapy for advanced disease allowed
* No prior chemotherapy within 4 weeks from treatment start (6 weeks in case of nitrosourea)
* No previous systemic corticosteroid therapy within 10 days
* Prior adjuvant treatment with IFN or other immunotherapy allowed
* Asymptomatic brain metastases allowed
* Measurable disease
* Prior treatment of brain metastases. In case stereotactic radiotherapy (or surgery) was not applicable, whole brain radiotherapy should have been performed
* Life expectancy >= 16 weeks
* ECOG performance status of 0 or 1
* Normal laboratory tests were required
* Negative screening tests for HIV, Hepatitis B, and Hepatitis C.
* Men and women, of and over 18 years old. Women of childbearing potential (WOCBP) must be using an adequate method of contraception to avoid pregnancy throughout the study and for up to 8 weeks after the study in such a manner that the risk of pregnancy is minimized.

Exclusion Criteria:

* Any malignancy from which the patient has been disease-free for less than 5 years, with the exception of adequately treated and cured basal or squamous cell skin cancer, superficial bladder cancer, carcinoma in situ of the cervix;
* Primary ocular or mucosal melanoma. Medical History and Concurrent Diseases
* Symptomatic brain metastases requiring immediate local intervention (radiotherapy (RT) and/or surgery)
* Autoimmune disease
* Any underlying medical condition, which in the opinion of the investigator, will make the administration of study drug hazardous or obscure the interpretation of adverse events, such as a condition associated with frequent diarrhea.

Prohibited Treatments and/or Therapies

* Concomitant therapy with any anti-cancer agent
* Immunosuppressive agents
* Any non-oncology vaccine therapy used for prevention of infectious diseases (for up to 1 month prior to or after any dose of study drug); surgery or radiotherapy ; other investigational anti-cancer therapies; or chronic use of systemic corticosteroids ;
* Previous treatment with other investigational products, including cancer immunotherapy, within 30 days;
* Previous enrollment in another clinical trial or prior treatment with a CD137 agonist or anti-CTLA-4 and/or fotemustine.

Sex and Reproductive Status

* WOCBP who are unwilling or unable to use an acceptable method to avoid pregnancy for the entire study period and for up to 8 weeks after the study;
* Women who are pregnant or breastfeeding;
* Women with a positive pregnancy test on enrollment or prior to investigational product administration;
* Sexually active fertile men not using effective birth control if their partners are WOCBP.

Other Exclusion Criteria

* Prisoners or subjects who are involuntarily incarcerated;
* Subjects who are compulsorily detained for treatment of either a psychiatric or physical illness.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 86 (Actual)
Dates: Start 2010-06; Primary Completion 2012-05 (Actual); Study Completion 2014-09 (Actual)

PRIMARY OUTCOMES:
The immune response disease control rate (irDCR) using the immune-related (ir) tumor response criteria of the combination of ipilimumab and fotemustine in patients with unresectable locally advanced or metastatic melanoma. | Weeks 24
  Immune-related Disease Control Rate (irDCR) is the proportion of treated subjects with a BOR of confirmed irCR, confirmed irPR or irSD.
  Tumor assessment (including determination of overall response at each tumor assessment and best overall response (BOR) taken over all tumor assessments prior to subsequent therapy is performed using the immune-related (ir) tumor response criteria.

SECONDARY OUTCOMES:
safety and feasibility of the combination of ipilimumab and fotemustine | 2 years
  A first clinical safety assessment will be performed to identify any early safety signals from ipilimumab given in combination with fotemustine at the first 18 treated patients. All subjects who receive at least 1 dose of study drug will be evaluable for safety parameters. Additionally, any occurrence of a SAE from time of consent forward will be reported.
Immune-related Major Durable Disease Control Rate (irMDDCR) | up to 24 weeks
  Immune-related Major Durable Disease Control Rate (irMDDCR) is the proportion of treated subjects with a duration of disease control of >= 24 weeks measured from Week 12, or (for those subjects with a confirmed irCR or confirmed irPR prior to Week 12) from the date of first overall response of irCR or irPR, until the date of irPD or death (whichever occurs first).
Immune-related Objective Response Rate (irORR) | Weeks 24
  Immune-related Objective Response Rate (irORR) is the proportion of treated subjects with a BOR of confirmed irCR or confirmed irPR.
Immune-related Time to Response (irTTR) | Weeks 24
  irTTR is defined as the time from first dosing date until the measurement criteria (using irRC) are first met for overall response of irPR or irCR (whichever status comes first, and provided it is subsequently confirmed).
Immune-related Progression-Free Survival (irPFS) | 2 years
  Immune-related Progression-Free Survival (irPFS) is defined as the time between the first dosing date and the date of irPD, or date of death, whichever occurs first. (ie, subjects who die without reported irPD will be considered to have progressed on the date of death).
Brain Progression-free Survival (Brain-PFS) | 2 years
  Brain Progression-free Survival (Brain-PFS) is defined as the time from first dosing date to the date of progression as per MRI of existing brain lesions, or of occurrence as per MRI of a new lesion located in the brain, or of death.
Overall Survival (OS) | 2 years
  Overall Survival (OS) is defined as the time from first dosing date until the date of death. For those subjects who have not died, OS will be censored at the recorded last date of subject contact, and for subjects with a missing recorded last date of contact, OS will be censored at the last date the subject was known to be alive.
  OS will be further described using the survival rate at one year, defined as the probability that a subject is alive at 1 and 2 years following first dose of study therapy and estimated via the Kaplan-Meier method.

CONTACTS AND LOCATIONS:
Overall Officials: Michele Maio, MD, PhD, Principal Investigator — Medical Oncology and Immunotherapy Unit, University Hospital of Siena
Locations (7):
- Italy (7):
  - National Institute for Cancer Research, Genoa
  - Immunotherapy and Somatic Cell Therapy Unit, Scientific Institute of Romagna, Meldola
  - European Institute of Oncology, Milan
  - Melanoma Unit, San Raffaele Hospital, Milan
  - Surgical Oncology, National Cancer Institute, Milan
  - Medical Oncology and Innovative Therapy, National Cancer Institute, Naples
  - Medical Oncology and Immunotherapy-University Hospital of Siena, Siena

REFERENCES:
- [Background] Robert C, Thomas L, Bondarenko I, O'Day S, Weber J, Garbe C, Lebbe C, Baurain JF, Testori A, Grob JJ, Davidson N, Richards J, Maio M, Hauschild A, Miller WH Jr, Gascon P, Lotem M, Harmankaya K, Ibrahim R, Francis S, Chen TT, Humphrey R, Hoos A, Wolchok JD. Ipilimumab plus dacarbazine for previously untreated metastatic melanoma. N Engl J Med. 2011 Jun 30;364(26):2517-26. doi: 10.1056/NEJMoa1104621. Epub 2011 Jun 5. PMID 21639810
- [Background] Hodi FS, O'Day SJ, McDermott DF, Weber RW, Sosman JA, Haanen JB, Gonzalez R, Robert C, Schadendorf D, Hassel JC, Akerley W, van den Eertwegh AJ, Lutzky J, Lorigan P, Vaubel JM, Linette GP, Hogg D, Ottensmeier CH, Lebbe C, Peschel C, Quirt I, Clark JI, Wolchok JD, Weber JS, Tian J, Yellin MJ, Nichol GM, Hoos A, Urba WJ. Improved survival with ipilimumab in patients with metastatic melanoma. N Engl J Med. 2010 Aug 19;363(8):711-23. doi: 10.1056/NEJMoa1003466. Epub 2010 Jun 5. PMID 20525992
- [Background] Avril MF, Aamdal S, Grob JJ, Hauschild A, Mohr P, Bonerandi JJ, Weichenthal M, Neuber K, Bieber T, Gilde K, Guillem Porta V, Fra J, Bonneterre J, Saiag P, Kamanabrou D, Pehamberger H, Sufliarsky J, Gonzalez Larriba JL, Scherrer A, Menu Y. Fotemustine compared with dacarbazine in patients with disseminated malignant melanoma: a phase III study. J Clin Oncol. 2004 Mar 15;22(6):1118-25. doi: 10.1200/JCO.2004.04.165. PMID 15020614
- [Background] Margolin K, Ernstoff MS, Hamid O, Lawrence D, McDermott D, Puzanov I, Wolchok JD, Clark JI, Sznol M, Logan TF, Richards J, Michener T, Balogh A, Heller KN, Hodi FS. Ipilimumab in patients with melanoma and brain metastases: an open-label, phase 2 trial. Lancet Oncol. 2012 May;13(5):459-65. doi: 10.1016/S1470-2045(12)70090-6. Epub 2012 Mar 27. PMID 22456429
- [Derived] Di Giacomo AM, Ascierto PA, Queirolo P, Pilla L, Ridolfi R, Santinami M, Testori A, Simeone E, Guidoboni M, Maurichi A, Orgiano L, Spadola G, Del Vecchio M, Danielli R, Calabro L, Annesi D, Giannarelli D, Maccalli C, Fonsatti E, Parmiani G, Maio M. Three-year follow-up of advanced melanoma patients who received ipilimumab plus fotemustine in the Italian Network for Tumor Biotherapy (NIBIT)-M1 phase II study. Ann Oncol. 2015 Apr;26(4):798-803. doi: 10.1093/annonc/mdu577. Epub 2014 Dec 23. PMID 25538176
- [Derived] Di Giacomo AM, Ascierto PA, Pilla L, Santinami M, Ferrucci PF, Giannarelli D, Marasco A, Rivoltini L, Simeone E, Nicoletti SV, Fonsatti E, Annesi D, Queirolo P, Testori A, Ridolfi R, Parmiani G, Maio M. Ipilimumab and fotemustine in patients with advanced melanoma (NIBIT-M1): an open-label, single-arm phase 2 trial. Lancet Oncol. 2012 Sep;13(9):879-86. doi: 10.1016/S1470-2045(12)70324-8. Epub 2012 Aug 13. PMID 22894884
- See also: Italian Network for Tumor Biotherapy (NIBIT) web-site, which will allow access to the diverse activities of the Network — http://www.nibit.org